CLINICAL TRIAL: NCT01364272
Title: Investigation of Diffusion Tensor Imaging Magnetic Resonance Imaging (DTI MRI) as a Correlate to Pain Relief and Facial Numbness in Patients Following Stereotactic Radiosurgical Rhizotomy for Trigeminal Neuralgia
Brief Title: Diffusion Tensor Imaging Magnetic Resonance Imaging (DTI MRI) as a Correlate to Pain Relief and Facial Numbness in Patients Following Stereotactic Radiosurgical Rhizotomy for Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Soltys, Associate Professor of Radiation Oncology, Stanford University
Other Study IDs: SU-05252011-7807; IRB 15136 (Other: Stanford IRB)
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Trigeminal neuralgia or tic douloureux is severe, often debilitating, facial pain that significantly impairs the patient's quality of life and health. Stereotactic radiosurgery has been shown to provide pain relief in majority of patients treated. However, a common side effect of radiosurgery is facial numbness. To better understand how radiosurgery can bring about pain relief and facial numbness, we are conducting a study in which brain MRI scans will be done following stereotactic radiosurgery to learn if there are any changes in the MRI scans that correlate with symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 years and older with typical trigeminal neuralgia, as determined by diagnostic criteria set by the International Headache Society, who are 1) intolerant of or refractory to medical management and 2) not candidates for or refusing a surgical micro-vascular decompression, will be evaluated for treatment with SRS.
* ECOG or Karnofsky Performance Status will not be employed, but patients must be sufficiently healthy to tolerate all study procedures.
* Patient must exhibit the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Exclusion criteria
* Patients who present with pre-existing facial numbness.
* Patients MRI contraindications (e.g., pacemaker or defibrillator, cochlear implant, brain aneurysm clip, etc.)
* Patients who have previously been treated with MVD.
* Patients who have previously had an ablative treatment, including prior SRS.
* Pediatric patients (age <18), pregnant women, and patients who are unable to give informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients age 18 years and older with typical trigeminal neuralgia, as determined by diagnostic criteria set by the International Headache Society, who was treated with SRS.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
DTI MRI findings | 6 months
  DTI MRI will be performed before and after radiosurgery to determine if there is a correlation between pain relief, facial numbness, and imaging changes.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Choi, Principal Investigator — Stanford University; Scott Soltys, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States